CLINICAL TRIAL: NCT03009851
Title: Testing an Occupation-Based Cultural Heritage Intervention in Long-Term Care Facilities
Brief Title: Testing the Effectiveness of an Occupation-based Cultural Intervention in Long-term Care
Acronym: OBCHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Retirement Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRF 2014-090
Record Dates: First submitted 2016-12-21; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Fragility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OBCHI (Experimental): This small group process intervention focuses upon the cultural heritage of the residents in LTC settings measuring quality of life, activity engagement and social participation.
  Interventions: Behavioral: OBCHI
- Control (No Intervention): The control group only received the typical activities conducted in LTC facilities.

INTERVENTIONS:
Behavioral: OBCHI — Occupation-based cultural heritage intervention emphasizing the cultural background of residents in LTC settings.
  Other Names: occupation-based cultural heritage intervention
  Arms: OBCHI

SUMMARY:
The goals of the proposed research were to:

1. describe the person and environment characteristics and activity patterns of residents in long-term care (LTC) facilities;
2. modify the evidence-based, occupation-based cultural heritage intervention (OBCHI) grounded on the results of Aim 1;
3. test the effectiveness of the OBCHI intended to facilitate adaptation to relocation into LTC facilities relative to a usual activities group;
4. determine the cost-effectiveness of the intervention conducted by in-house staff compared to the control group; and
5. examine person and environment factors as potential moderators of the relationship between treatment condition and adaptation outcomes.

DETAILED DESCRIPTION:
Specific Aims

Primary Aims

1. Describe the person and environment characteristics and activity patterns of residents in LTC facilities.
2. Modify the OBCHI grounded on the evidence-based results of Aim 1 specific to these facilities and residents.
3. Test the effectiveness of the OBCHI conducted by activity department staff, relative to usual activities, as measured by quality of life, activity engagement, and social participation.

   H1a-c: Those receiving OBCHI will have significantly greater improvement in

   a) quality of life, b) activity engagement, and c) social participation at post-intervention relative to those receiving usual activities.

   H2a-c: Those receiving OBCHI will have greater maintenance of improvements in a) quality of life, b) activity engagement, and c) social participation at 1-month follow-up, relative to those receiving usual activities.
4. Determine the cost-effectiveness of the intervention in terms of quality adjusted life year (QALY) and other health factors.

   H3: When OBCHI is proven to be more effective in promoting quality of life than usual activities, the investigators will expect the OBCHI to produce a higher QALY at a lower cost per QALY.

   H4: Between these two mutually exclusive treatments, the OBCHI intervention will be more efficient (more effective and less costly) or cost saving with a negative incremental cost-effectiveness ratio (ICER) when compared to those receiving usual activities.

   Exploratory Aim
5. Examine person characteristics (i.e. cultural heritage, life experiences social support, resilience, depression, and resident demographics [age, gender, ethnicity]) and select environment characteristics (i.e., participant perceptions of the intervention and facility) as potential moderators of the relationship between treatment condition (OBCHI versus usual care) and change in adaptation outcomes from pre- to post-intervention.

Table 1. Timeline of Person/Environment Factors, Outcomes and Tools

Person Characteristics Tools Baseline 1 wk. post 1 m. follow-up

Cognitive Screen SPMSQ x

Life Experience Interview x

Social Support Yesterday Interview x x x

Resilience Resilience Scale x

Depression GDS-15 x x x

Environment Characteristics

LTC Facility Setting Site Demographics x

Resident Perceptions SCES x x x Intervention Evaluation (midway) x

Staff Perceptions Questionnaire x x

Outcomes

QoL QOLI/SF-12 x x x

Cost Effectiveness SF-12 x x x

Activity Engagement and Social Participation Yesterday Interview x x x

Significance

As the need for LTC increases with the steady growth of older adults, relocation into residential settings will grow. About 70 percent of persons over 65 will require spending time in LTC services, with 40 percent requiring nursing home care for a period of time. Relocation is moving from one permanent home to another permanent home which is sometimes precipitated by an illness and considered a significant life event. Skinner noted a forced relocation could have disturbing effects upon the elderly including loss of social and community connections. However, even with a planned relocation, encountering this new and unfamiliar environment requires the older person to rethink the ways in which his or her life will differ with adjustment duration of a few weeks to several years. Many factors determine the ways in which this 'new life' will evolve including: past adaptive strategies and life experiences, family support systems, socioeconomic resources, and cultural values.

Moving from a familiar environment to an unfamiliar one involves adaptation, regardless of age. Adaptation is a process involving interaction between the person and environment. Indicators of successful adaptation to LTC have included: developing a sense of identity and place, having care needs met, knowing and being known to other residents, maintaining or developing social networks, continuity of lifestyle, and maintaining control over life situations. As defined for this study, adaptation is a normal process by which a person encounters a perceived challenge in the environment and is able to successfully manage that challenge as measured by increased quality of life, activity engagement and social participation. Central to adaptation is the cultural heritage that an individual brings to the LTC facility upon relocation. Because culture is the learned beliefs, values, customs, actions, communication, and life ways of an individual, it can be expected to permeate all aspects of life in a residential facility. Attention to an individual's cultural heritage has begun to make in-roads to the daily life routines encountered in these facilities.

Acknowledgement of the resident's culture is a major contributing factor to his/her quality of life (QOL). However, QOL is a complex construct and has been used synonymously with terms like well-being, life satisfaction, and functional health. Lawton asserted that QOL is a collection of dimensions comprised of both objective and subjective factors which may include all or some of the following: behavioral competence, objective environment, perceived QOL, psychological well-being, and health-related status. Other factors associated with QOL include: interaction with family and friends, personal qualities, room and meal items, number of health problems, staff-resident ratios and continuity of care. These findings attest to the importance of a person-environment 'match' when QOL issues for residents are considered.

Incorporating meaningful activity and social connections into the lives of elders that have been circumscribed by illness and disability is particularly important to QOL. Gerontological literature concerning the activities of elders has concentrated upon personal care and instrumental activities and how they contribute to health and functional status. These obligatory tasks are essential to one's survival, but perhaps even more significant to an elder's well-being are those discretionary activities involving social and meaningful occupations; such findings support the proposition that activity and social support systems are important in mediating the impact of illness on well-being.

In summary, the relationship of relocation, culture, adaptation, QOL, activity engagement, and social participation is reflected in outcomes where failure to provide culturally competent and culturally sensitive care have occurred. With increasing diversity of the US population, practitioners are challenged to deliver culturally competent services and to improve the QOL for diverse LTC residents.

ELIGIBILITY:
Inclusion Criteria:

* English speaking, less than one year from admission, cognitive level of 4/5 on SPMSQ

Exclusion Criteria:

* non English speaking, more than one year in LTC, and less than cut off score on SPMSQ

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Change is being assessed at baseline, 1 week and 1 month follow up
  QOLNH by Ferran

SECONDARY OUTCOMES:
SF-12 | Change is being assessed at baseline, 1 week and 1 month follow up
  Measurement of general health

CONTACTS AND LOCATIONS:
Overall Officials: Donna Tilley, PhD, Study Director — Texas Woman's University
Locations (1):
- Texas Woman's University, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be presented without names and by treatment and/or control group. Information may include: gender, age, ethnicity, education level, and/or scores from the outcome measures. This information will be shared via publications and professional presentations.
  The IRB is currently approved and continues to be renewed on a yearly basis. Contact the PI for further information.